CLINICAL TRIAL: NCT05303753
Title: An Exploratory Study on the Effect of Fermented Dairy Protein With Prebiotic Fiber in Athletes
Brief Title: Protein-Prebiotic Wellbeing Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00014399
Record Dates: First submitted 2022-02-14; First posted 2022-03-31 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Digestive Health; Quality of Life
Keywords: Participants; Healthy subjects; Athlete; Women; Men; Fermented Dairy; Prebiotics; Gut microbiota; Self-reported; GI tract; Diet; Sleep
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: Modifying diet by adding a fermented dairy protein with prebiotic fiber
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Other): During a 3-week baseline period, participants with self-reported GI complaints consume their own protein supplement that they use for recovery purposes after exercise, followed by a 3-week intervention period in which they maintain usage of their own product, but replace a part of this product with a fermented dairy protein with prebiotic fiber. An additional reference group of athletes without self-reported GI complaints will also be followed during a 3-week period in which they consume their own protein supplement that they use for recovery purposes after exercise.
  Interventions: Other: fermented dairy protein with prebiotic fiber

INTERVENTIONS:
Other: fermented dairy protein with prebiotic fiber — During the intervention period, the participant will consume a new product and will reduce the amount of protein in their normal diet reflecting the protein content of the new product.

SUMMARY:
Healthy participants with self-reported GI complaints will consume the protein supplement that they normally use for recovery purposes after exercise during a 3-week baseline period, followed by a 3-week intervention period in which they maintain usage of their product, but replace a part of this product with a fermented dairy protein with prebiotic fiber. In addition, a group of healthy participants without self-reported GI complaints will serve as a reference group by consuming the protein supplement that they normally use for recovery purposes after exercise during a 3-week period.

DETAILED DESCRIPTION:
A substantial number of athletes suffer from gastro-intestinal problems, which may impair performance and/or subsequent recovery. Also, gut barrier integrity is impaired with high-intensity training. Emerging studies are showing a positive correlation between the gut microbiome and muscle function, athletic performance, body composition, and natural energy levels. This study will perform an exploratory analysis of the well-being and digestive health of well-trained athletes, and assess the potential effect of fermented dairy protein with prebiotic fiber on these parameters.

Question 1: Does the 3-week supplementation of a fermented dairy protein with prebiotic fiber affect the self-reported digestive comfort compared to a 3-week baseline period? And additionally, will the quality of life (self-reported general well-being and states of mood) change with the use of this type of product?

Question 2: Does the 3-week supplementation of a fermented dairy protein with prebiotic fiber show an alteration in gut microbiota in comparison to a 3-week baseline period, while dietary intake remains unaffected?

Question 3: How is the 3-week supplementation of a fermented dairy protein with prebiotic fiber experienced by the participants (taste and concept liking)?

Question 4: Is there a difference in baseline gut microbiota between athletes with and athletes without self-reported GI complaints.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects living in Arizona in the USA
* Women/Men aged between 18-35 years
* Serious athletes (exercise at least 3 x per week)
* With or without GI tract issues due to sport or protein/diet intake
* 18.5 ≤ BMI ≤ 40 kg/m2
* No physical limitations (i.e. able to perform all activities associated with daily living in an independent manner).
* Use of a protein supplement or sports food after at least one training per day 3 x per week
* Willing to slightly increase their protein supplement intake during the intervention phase for 21 consecutive days
* Stable weight during the last 4 weeks, without a focus on body weight reduction through limiting caloric intake
* Written informed consent

Exclusion Criteria:

* Daily use of (sport) supplements containing probiotics and/or prebiotics
* Smoking
* Self-reported cow's milk protein allergy
* Clinical lactose intolerance
* Clinical milk protein allergy
* House dust mite allergy
* Diagnosed GI tract disorders or diseases
* Musculoskeletal disorders
* Metabolic disorders (such as diabetes)
* Use of any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescribed acne medications).
* Chronic use of gastric acid-suppressing medication or anti-coagulants
* Use of antibiotics or anti-inflammatory medication the past 2 weeks
* Blood donation in the past 2 months
* Pregnant/lactating women
* Athletes should not aim to lose body weight by reducing energy intake during the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants can identify as: Male, Female, Non-binary/third gender, or as: Prefer not to say.
Enrollment: 98 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Change in self-reported digestive comfort | Baseline (day 0), after 21 days and after 42 days.
  Gastrointestinal Symptoms Rating Scores (GSRS-score: Average of all 5 sub-scores)
Change in daily self-reported digestive comfort | Study period covering day 1 to day 21 compared to day 22-42.
  Daily variation of GI complaints (averaged itemized score 1-10)

SECONDARY OUTCOMES:
Change in self-reported general wellbeing - Physical Health | Baseline (day 0), after 21 days and after 42 days.
  Reported as physical wellbeing (Physical Health Questionnaire, PHX - average score 1-7 based on 14 items)
Change in self-reported general wellbeing - Psychological Distress | Baseline (day 0), after 21 days and after 42 days.
  Reported as psychological distress (mental distress, K6 scale - average score 0-24).
Change in participants microbiota composition of fecal samples | Baseline (day 0), after 21 days and after 42 days.
  16s microbial profiling
Change in dietary intake | Baseline (day 0), after 21 days and after 42 days.
  24-hour dietary recalls (food group intake, energy and macro- and micronutrient)
Chane in self-reported states of mood | Baseline (day 0), after 21 days and after 42 days.
  Profile of Mood States (POMS)

OTHER OUTCOMES:
Change in food composition and diet quality | Baseline (day 0), after 21 days and after 42 days.
  Rapid eating assessment in participants (REAP)
Change in product experience | Baseline (day 0), days 22, 23, 29, 36, 43.
  Question about product experience (taste and concept liking)

CONTACTS AND LOCATIONS:
Overall Officials: Floris Wardenaar, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No